CLINICAL TRIAL: NCT01233622
Title: A Multi-center, Randomized, Double-blind Placebo Controlled Study to Evaluate the Efficacy and Safety of 24 Weeks Treatment With Vildagliptin 50 mg Bid as add-on Therapy to Metformin Plus Glimepiride in Patients With Type 2 Diabetes
Brief Title: Safety and Efficacy of Galvus as add-on Therapy to Metformin Plus Glimepiride
Acronym: Vildagliptin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A23152; EudraCT 2010-021097-11
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (metformin + glimepiride) (Experimental)
  Interventions: Drug: Vildagliptin
- Placebo (metformin + glimepiride) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin (metformin + glimepiride)
Drug: Placebo
  Arms: Placebo (metformin + glimepiride)

SUMMARY:
This study will evaluate the efficacy and safety of vildagliptin 50 mg bid as add-on therapy to metformin plus glimepiride in patients with Type 2 Diabetes (T2D).

ELIGIBILITY:
Inclusion criteria

* Confirmed diagnosis of T2DM by standard criteria.
* Treatment with oral anti-diabetic therapy, on stable dose for at least 12 weeks prior to the screening visit. Acceptable background anti-diabetic therapy includes: metformin (≥ 1500 mg) as monotherapy or in combination with SU, TZDs, or glinides
* Age: ≥18 to ≤ 80 years
* HbA1c of ≥ 7.5 and ≤ 11.0%
* Body Mass Index (BMI) ≥22 to ≤45 kg/m2

Exclusion criteria:

* FPG ≥ 270 mg/dL (≥ 15.0 mmol/L)
* Acute metabolic diabetes complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months
* Any of following within past 6 months: Myocardial infarction, TIA or stroke, coronary artery bypass surgery or percutaneous coronary intervention
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Acute infections which may affect blood glucose control within 4 weeks prior to screening Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
HbA1c Reduction | 24 weeks

SECONDARY OUTCOMES:
FPG reduction | 24 weeks
Safety and tolerability-frequency of treatment emergent adverse events (incl. overall Aes, SAEs, death, Aes leading ot study discontinuation or study drug interruption, pre-specified potential AEs) | 24 weeks
Responder Rate | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- Australia (4):
  - Novartis Investigative Site, Box Hill
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Parkville
  - Novartis Investigative Site, St Leonards
- Germany (8):
  - Novartis Investigative Site, Anderbeck
  - Novartis Investigative Site #1, Berlin
  - Novartis Investigative Site #2, Berlin
  - Novartis Investigative Site #3, Berlin
  - Novartis Investigative Site #4, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Sangerhausen
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Érd
  - Novartis Investigative Site, Törökbálint
- Italy (8):
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Cosenza
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site #1, Roma
  - Novartis Investigative Site #2, Roma
  - Novartis Investigative Site, Torino
- Mexico (15):
  - Novartis Investigative Site #1, Aguascalientes
  - Novartis Investigative Site #2, Aguascalientes
  - Novartis Investigative Site #3, Aguascalientes
  - Novartis Investigative Site #1, Durango
  - Novartis Investigative Site #2, Durango
  - Novartis Investigative Site #3, Durango
  - Novartis Investigative Site #1, Guadalajara
  - Novartis Investigative Site #2, Guadalajara
  - Novartis Investigative Site #3, Guadalajara
  - Novartis Investigative Site #4, Guadalajara
  - Novartis Investigative Site #5, Guadalajara
  - Novartis Investigative Site, México
  - Novartis Investigative Site #1, Pachuca
  - Novartis Investigative Site #2, Pachuca
  - Novartis Investigative Site #3, Pachuca
- Philippines (3):
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site #1, Quezon City
  - Novartis Investigative Site #2, Quezon City
- Romania (5):
  - Novartis Investigative Site, Alba Iulia
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site #1, Oradea
  - Novartis Investigative Site #2, Oradea
  - Novartis Investigative Site, Târgu Mureş
- South Korea (5):
  - Novartis Investigative Site, Bundang
  - Novartis Investigative Site #1, Seoul
  - Novartis Investigative Site #2, Seoul
  - Novartis Investigative Site #3, Seoul
  - Novartis Investigative Site, Suwon
- Taiwan (4):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Yongkang District

REFERENCES:
- [Result] Lukashevich V, Del Prato S, Araga M, Kothny W. Efficacy and safety of vildagliptin in patients with type 2 diabetes mellitus inadequately controlled with dual combination of metformin and sulphonylurea. Diabetes Obes Metab. 2014 May;16(5):403-9. doi: 10.1111/dom.12229. Epub 2013 Dec 2. PMID 24199686